CLINICAL TRIAL: NCT03639285
Title: Natural History, Diagnosis, and Outcomes for Leukodystrophies
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Josh Bonkowsky, Professor, Principal Investigator, University of Utah
Other Study IDs: 00019596
Record Dates: First submitted 2018-07-28; First posted 2018-08-21 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Leukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Patients have the option to have a DNA sample or cell line sample biobanked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goals of this protocol is to diagnose, care for, and understand the clinical histories and outcomes of people with leukodystrophies.

DETAILED DESCRIPTION:
Inherited leukodystrophies affect close to 1 in 7500 children with mortality greater than 30%. Affected patients face additional serious medical complications including epilepsy, developmental regression, and intellectual disabilities. Diagnosis is difficult and requires the assistance of a specialist. Finally, identifying treatments and improving outcomes is complex.

The Western Leukodystrophy Project, which is part of the University of Utah and of Primary Children's Hospital, and which is a certified Leukodystrophy Care Network Center, provides a specialized resource for patients with leukodystrophies.

This clinical study assists with diagnosis of leukodystrophies; suggesting treatment options and implementing care guidelines, and improving outcomes for all patients by understanding the clinical histories and outcomes of affected patients..

ELIGIBILITY:
Inclusion Criteria:

* evidence by clinical exam, radiological findings, and/or testing, of an inherited leukodystrophy.
* be able to travel to the leukodystrophy clinic (at Primary Children's Hospital, Salt Lake City, Utah);
* be able to tolerate a general physical exam, and a neurological exam.

Exclusion Criteria:

* unable to be evaluated at the University of Utah Hospital or Primary Children's Hospital;
* refusal to sign study consent form;
* evidence or finding of another non-genetic cause of their condition;
* Persons with known white matter disease or lesions related to: birth injury or prenatal injury, multiple sclerosis, trauma, infection, immunization, or post-infectious effects (e.g. ADEM- acute disseminated encephalomyelitis), metabolic disturbance (e.g. Central pontine myelinolysis), neoplasms, primary rheumatologic diseases (e.g. Systemic lupus erythematosis), stroke, hypoxic-ischemic injury, drug or toxin effect, seizures, or endocrine disturbance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person with an apparent inherited disease of white matter (except as excluded by the exclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-01-19 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Determine rates of morbidity

SECONDARY OUTCOMES:
Hospitalizations | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Number of hospitalizations
MRI of the brain | Participants will be followed for the duration of the study (up to 20 years), with an MRI performed at presentation and then repeated on average once every 5 years
  Perform brain MRI to evaluate changes due to a leukodystrophy
Diagnosis | Participants will be tested at presentation, and then re-tested for the duration of the study (up to 20 years), with re-testing on average of once per three years
  Using sequencing to establish a genetic diagnosis
Response to bone marrow transplant | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate neurological changes due to leukodystrophy and response following a bone marrow
Spasticity complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate spasticity complications defined by the presence of increased tone (spasticity)
Respiratory complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate respiratory complications defined by the need for supplemental oxygen
Hypotonia complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate hypotonia complications defined by the presence of hypotonia
Bulbar complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate bulbar complications defined by the presence of swallowing difficulties
Cerebellar complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate cerebellar complications defined by the presence of ataxia or coordination problems
Language complications | Participants will be followed for the duration of the study (up to 20 years), with checks on average of once per year
  Evaluate language complications defined by language impairment below age norms

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Children's Hospital, Salt Lake City, Utah, United States